CLINICAL TRIAL: NCT02139332
Title: A Primary Prevention Trial to Strengthen Child Attachment in a Native Community
Acronym: FPT PFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Cathryn Booth-LaForce, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00010153; 5R01NR014153-05 (NIH)
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Parent-child Interaction
Keywords: Attachment theory; Parent- child relationship; Child mental health; Behavioral health
MeSH Terms: interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resource & Referral group (Active Comparator): Individuals randomized to the control group will receive a resource & Referral service immediately after their baseline research visit.
  Interventions: Behavioral: Resource & Referral Group
- PFR Group (Experimental): Individuals randomized to the Immediate group will receive the intervention program immediately after completing the baseline assessment.
  Interventions: Behavioral: PFR Group

INTERVENTIONS:
Behavioral: PFR Group — The intervention consists of delivering the Promoting First Relationship (PFR) program. PFR comprises 10 sessions and lasts approximately 12 weeks. Each session begins with a brief discussion and education on the target topic for that week . Then 20 minutes is spent on video recording a structured interaction between the caregiver and child or viewing the previous session's recording and engaging in reflective discussion about successful caregiving strategies and child's response to caregiver behavior (alternating weeks). Trained PFR specialists who are community members use the 5 "consultation strategies," labeled Joining, Positive Feedback, Instructive Feedback, Reflective Questions and Comments, and Instruction with Handouts.
  Arms: PFR Group
Behavioral: Resource & Referral Group — The Resource & Referral program consists of 1) an initial needs assessment to determine if the enrolled family has any unmet needs (housing, financial, health, mental health, etc…), 2) a tailored resource and referral packet will be mailed to the participant with the most important referrals marked, 3) a follow-up call will be made two weeks after mailing the packet to verify that the participant has received it, and 4) a second follow-up call will be made three months after the initial session, to assess types of services actually received, barriers to receiving services, and reassessing resources needed and providing additional referrals if needed.
  Arms: Resource & Referral group

SUMMARY:
The purpose of this study is to to conduct a randomized controlled trial comparing an intervention group and a control group to evaluate the feasibility of the Promoting First Relationships method in an American Indian community through their tribal Health Promotion program, and to assess the efficacy of the method in this community.

ELIGIBILITY:
Inclusion Criteria:

1. Primary caregiver for a child aged 10 to 30 months
2. Caregiver lives with the child full time for the past three months and plans to continue for at least 6 more months.
3. Child is an American Indian or Alaska Native living on or near the Tribe's reservation.
4. Caregiver has telephone access
5. Caregiver is willing to have researchers come to their house
6. Caregiver is English speaking
7. Caregiver is willing to participate in a home-visiting program which includes video-recorded sessions of caregivers and their children playing

Exclusion Criteria: Caregiver is

1. Hospitalized or imprisoned
2. Living in a Treatment facility or shelter
3. Unable to give consent
4. Live in a household that already has a dyad enrolled in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of caregiver-child interactions from baseline at 3 months and 6 months | Baseline, 3-month and 6-month follow-ups
  We are using the Nursing Child Assessment Satellite Training Teaching Scales to assess quality of caregiver-child interactions. Caregivers select an activity that their child cannot perform, such as drawing, and spend up to 5 minutes teaching this activity to the child. The interaction is video-recorded and coded for the caregiver's sensitivity to cues, response to distress, and fostering of social, emotional, and cognitive growth, as well as for the child's clarity of cues and responsiveness to the caregiver.

SECONDARY OUTCOMES:
Change in Caregiver helplessness from baseline at 3 months and 6 months | Baseline, 3-month and 6-month follow-ups
  Caregiver helplessness is measured by the Caregiving Helplessness Questionnaire, comprising 45 items specific to interactions with the child. We evaluate 2 subscales for this study: Mother-Child Frightened and Mother Helplessness ("mother" is changed to "caregiver")
Change in Caregiver stress from baseline at 3 months and 6 months | Baseline, 3-month and 6-month follow-ups
  Caregiver stress is measured by the Parenting Stress Index/Short Form, a 36-item questionnaire with 3 subscales: caregiver distress, caregiver-child dysfunctional interaction, and difficult child.
Change in Child Social-emotional Competence from baseline at 3 months and 6 months | Baseline, 3-month and 6-month follow ups
  Children's social-emotional competencies are measured with the Infant-Toddler Social Emotional Assessment, a caregiver-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cathryn Booth-LaForce, PhD, Principal Investigator — University of Washington
Locations (1):
- MBIRI, Eagle Butte, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oxford M, Booth-LaForce C, Echo-Hawk A, Madesclaire O, Parrish L, Widner M, Petras A, Abrahamson-Richards T, Nelson K, Buchwald D; CATCH Project Team. Promoting First Relationships(R): Implementing a Home Visiting Research Program in Two American Indian Communities. Can J Nurs Res. 2020 Jun;52(2):149-156. doi: 10.1177/0844562120914424. Epub 2020 Mar 26. PMID 32216455
- [Derived] Booth-LaForce C, Oxford ML, O'Leary R, Rees J, Petras A, Buchwald DS. Implementation fidelity of the Promoting First Relationships intervention program in a Native community. Transl Behav Med. 2023 Jan 20;13(1):34-41. doi: 10.1093/tbm/ibac060. PMID 36227860